CLINICAL TRIAL: NCT05132894
Title: An Osteopathic Assessment of Lower Extremity Somatic Dysfunction in Runners
Status: Completed | Type: Observational
Sponsor: The Touro College and University System (Other)
Responsible Party: Principal Investigator, Abbey Santanello, Principal Investigator, OMS-IV, The Touro College and University System
Other Study IDs: 001
Record Dates: First submitted 2021-09-13; First posted 2021-11-24 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Somatic Dysfunction of Sacral Region; Somatic Dysfunction of Both Sacroiliac Joints; Somatic Dysfunction of Bilateral Lower Extremities
Keywords: somatic dysfunction; runners; osteopathic; osteopathic assessment; lower extremity; lower extremity somatic dysfunction; running injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Novice Runners: 1-5 miles / week 18+ yo
  Interventions: Other: Osteopathic Assessment
- Moderate Runners: 6-15 miles / week 18+ yo
  Interventions: Other: Osteopathic Assessment
- Advanced Runners: 16+ miles / week 18+ yo
  Interventions: Other: Osteopathic Assessment

INTERVENTIONS:
Other: Osteopathic Assessment — As osteopathic structural exam will be performed to assessment somatic dysfunctions of the lower extremities.

SUMMARY:
Runners often experience acute/chronic pain due to pre-existing structural somatic dysfunction and/or acquired various overuse injuries of the lower extremity, specifically affecting the ligaments, tendons, muscles and bones. Common structural and function dysfunctions include but are not limited to patellofemoral pain syndrome (PFPS), Achilles tendonitis, iliotibial band syndrome (ITBS), ligamentous and muscle tears, muscle sprains/strains, stress fractures, pes planus, plantar fasciitis, and shin splints.

The purpose of this study is to assess the correlation between acute and chronic pain, overuse injuries, and observational and palpatory findings upon evaluation. With an understanding of the common trends of somatic dysfunctions and etiology of the pain/injury, modified regimen/routine and improved treatment plans can be developed and recommended for runners to better rehabilitate, minimize relapse and reduce compensatory injuries. No medical or osteopathic treatment will be provided.

ELIGIBILITY:
Inclusion Criteria:

* Self-proclaimed runners that run at least 1 mile per week consistently
* Minimum 18 years old

Exclusion Criteria:

* Non-runners
* Inconsistent runners, do not log at least 1 mile weekly

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population includes any adult-aged males and females that are self-proclaimed runners confirming that they run at least 1 mile per week. The runners will be categorized based on the quantity of miles run weekly.
  The sampling method is non-probability for convenience to easily gather data.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2021-11-20 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-02-20 (Actual)

PRIMARY OUTCOMES:
Structural exam to determine type of Lower Extremity Somatic Dysfunctions in participants | up to 8 weeks
  Osteopathic Structural Exam to assess changes to muscles, bones, bursae, and ligaments
Questionnaire to analyze data on runners' background/history | up to 8 weeks
  Questionnaire to learn about runners' background

CONTACTS AND LOCATIONS:
Locations (1):
- Touro College of Osteopathic Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Amount of Running and Association With Risk of All-Cause, Cardiovascular, and Cancer Mortality — https://www.practiceupdate.com/content/amount-of-running-and-association-with-risk-of-all-cause-cardiovascular-and-cancer-mortality/92176/37/6/1?elsca1=TrendMD_CPA&origin=b3610ec5cf201fa8306d1680c13278de
- See also: Is running associated with a lower risk of all-cause, cardiovascular and cancer mortality, and is the more the better? A systematic review and meta-analysis — https://bjsm.bmj.com/content/early/2019/09/25/bjsports-2018-100493
- See also: Controlled trial to compare the Achilles tendon load during running in flatfeet participants using a customized arch support orthoses vs an orthotic heel lift. — https://doi.org/10.1186/s12891-019-2898-0
- See also: Overuse Injury: The Result of Pathologically Altered Myofascial Force Transmission? — https://journals.lww.com/acsm-essr/Abstract/2019/10000/Overuse_Injury__The_Result_of_Pathologically.6.aspx
- See also: Diseases and overuse injuries of the lower extremities in long distance runners — https://europepmc.org/article/MED/28236094
- See also: Incidence of Running-Related Injuries Per 1000 h of running in Different Types of Runners: A Systematic Review and Meta-Analysis — https://link.springer.com/article/10.1007/s40279-015-0333-8
- See also: Lower Extremity Injuries in Runners — https://link.springer.com/article/10.2165/00007256-199213010-00005